CLINICAL TRIAL: NCT03775382
Title: Mechanisms of Impaired Brain Blood Flow With Aging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Responsible Party: Principal Investigator, Christopher Martens, Assistant Professor, University of Delaware
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: Martens - 1138735
Record Dates: First submitted 2018-12-06; First posted 2018-12-13 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Aging
MeSH Terms: interventions — Ascorbic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Normal saline will be infused by the research nurse into an antecubital vein using an IV infusion pump.
  Interventions: Other: Normal Saline
- Ascorbic Acid (Active Comparator): Ascorbic acid will be measured into sterile syringes by the research nurse and infused into an antecubital vein using a IV infusion pump beginning with a priming bolus of 0.06 g Ascorbic Acid per kg fat-free mass dissolved in 100 ml of saline or lactated ringers followed by a "drip-infusion" of 0.02 g Ascorbic Acid per kg fat-free mass dissolved in 30 ml of saline.
  Interventions: Other: Ascorbic Acid

INTERVENTIONS:
Other: Ascorbic Acid — Ascorbic acid will be infused into an antecubital vein using a IV infusion pump beginning with a priming bolus of 0.06 g Ascorbic Acid per kg fat-free mass dissolved in 100 ml of saline followed by a "drip-infusion" of 0.02 g Ascorbic Acid per kg fat-free mass dissolved in 30 ml of saline.
  Other Names: Vitamin C
  Arms: Ascorbic Acid
Other: Normal Saline — Normal saline will be infused by the research nurse into an antecubital vein using an IV infusion pump.
  Arms: Placebo

SUMMARY:
Aging is the primary risk factor for Alzheimer's disease (AD), which is a rapidly growing public health concern. Understanding the mechanisms of normal brain aging may provide insight into the factors linking advancing age to increased risk for AD and thereby lead to new therapeutic targets for preventing or slowing AD progression. Cardiovascular changes, including impaired cerebrovascular function, occur with aging and may increase risk for AD; however, the mechanisms by which cerebrovascular function becomes impaired in older adults are incompletely understood. The overall goal of this project is to examine potential mechanisms of age-related declines in cerebrovascular function in humans. The investigators hypothesize that brain macro-vascular endothelial dysfunction, secondary to oxidative stress, plays an important role in mediating age-related changes in brain blood flow and cerebrovascular reactivity. The results of this pilot study have the potential to identify novel targets of cerebrovascular aging and will help guide the design of future clinical trials aimed at improving cerebral blood flow in older adults.

ELIGIBILITY:
Inclusion Criteria:

* 18-29 or 55-79 years old

Exclusion Criteria:

* Pregnancy or breastfeeding;
* Blood chemistries indicative of abnormal renal, liver, thyroid and adrenal function (i.e., outside of normal reference range); estimated glomerular filtration rate using the MDRD prediction equation must be >60 ml/min/1.73 m2;
* Abnormal blood chemistry that is clinically relevant or any blood chemistry marker that is +/-2.5x the upper or lower limit;
* Lack of a suitable temporal window for cerebrovascular assessments;
* Current smoking;
* Chronic clinical diseases (e.g., coronary artery, peripheral artery, or cerebrovascular diseases, diabetes, chronic kidney disease, COPD);
* Major psychiatric disorder (e.g. Alzheimer's disease or other form of dementia, schizophrenia, bipolar disorder, major depression within past two years);
* Neurological or autoimmune conditions affecting cognition (e.g. Parkinson's disease, epilepsy, multiple sclerosis, head trauma with loss of consciousness greater than 30 min, large vessel infarct);
* Current medication use likely to affect CNS functions (e.g. long active benzodiazepines);
* Having past or present alcohol dependence or abuse, as defined by the American Psychiatry Association, Diagnostic and Statistical Manual of Mental Disorders;
* Body mass index (BMI) >40 kg/m2 (FMD measurements can be inaccurate in severely obese patients).

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in internal carotid artery (ICA) diameter after acute infusion of the antioxidant ascorbic acid | Change from baseline to 30 minutes post-infusion
  Cerebrovascular reactivity to hypercapnia

SECONDARY OUTCOMES:
Change from baseline in middle cerebral artery (MCA) diameter after acute infusion of the antioxidant ascorbic acid | Change from baseline to 30 minutes post-infusion
  Cerebrovascular reactivity to hypercapnia

CONTACTS AND LOCATIONS:
Overall Officials: Christopher R Martens, Ph.D., Principal Investigator — University of Delaware
Locations (1):
- Neurovascular Aging Laboratory, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No